CLINICAL TRIAL: NCT04718883
Title: A Phase II Open-Label, Single-Arm, Multicenter Study of JWCAR029, CD19-targeted Chimeric Antigen Receptor (CAR) T Cells for Relapsed and Refractory (R/R) Mantle Cell Lymphoma
Brief Title: CD19-targeted CAR T Cells for Relapsed and Refractory (R/R) Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029-005
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Mantle Cell Lymphoma
Keywords: JWCAR029; B-Cell Malignancies; Non-Hodgkin lymphoma; CAR T cells; Chimeric antigen receptor; Relapsed/Refractory; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Recurrence | interventions — Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR029 treatment (Experimental): JWCAR029 be administrated at dose level: 1 x 10^8 CAR+T cells
  Interventions: Biological: CD19-targeted Chimeric Antigen Receptor (CAR) T Cells

INTERVENTIONS:
Biological: CD19-targeted Chimeric Antigen Receptor (CAR) T Cells — JWCAR029 will be administered at dose level: 1 x 10^8 CAR+T cells

SUMMARY:
This is a phase II, open-label, single-arm, multicenter study to assess the efficacy and safety of JWCAR029 in adult R/R Mantle Cell Lymphoma subjects in China.

DETAILED DESCRIPTION:
This is a phase II, open-label, single-arm, multicenter study conducted in adult subjects with relapsed and refractory (R/R) mantle cell lymphoma (MCL) in China to evaluate the safety, efficacy, pharmacokinetics(PK), pharmacodynamics(PD) of JWCAR029 and immune response after JWCAR029 treatment.

R/R MCL patients will be enrolled in dose level of 1.0 x 10^8 CAR+ T cells. All subjects will be followed for 5 years following JWCAR029 infusion.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* Sign on the informed consent;
* Subject must have histologically confirmed mantle cell lymphoma;
* Relapsed/refractory patients;
* Subjects have accessible PET-positive lesion and have measurable CT-positive lesion according to Lugano Classification;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Expected survival is greater than 12 weeks;
* Adequate organ function;
* Adequate vascular access for leukapheresis procedure;
* Subjects who have previously received CD19 targeted therapy must confirm that lymphoma lesions still express CD19;
* Women of childbearing potential must agree to use highly effective methods of contraception for 1 year after the last dose of JWCAR029;
* Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 1 year after the last dose of JWCAR029.

Exclusion Criteria:

* Central nervous system (CNS) only involvement by malignancy or primary CNS lymphoma;
* History of another primary malignancy that has not been in remission for at least 2 years;
* Subjects has HBV, HCV, HIV or syphilis infection at the time of screening;
* Deep venous thrombosis (DVT)/Pulmonary embolism (PE), or DVT/PE requires anti-coagulation within 3 months prior to signing the ICF;
* Subjects with uncontrolled systemic fungal, bacterial, viral or other infection;
* Presence of acute or chronic graft-versus-host disease (GVHD);
* History of any serious cardiovascular disease or presence of clinically relevant CNS pathology;
* Pregnant or nursing women;
* Subjects using of any chemotherapy, corticosteriod, experiment agents, GVHD therapies, radiation or any other therapies for lymphoma must go through a specific wash-out period before leukapheresis;
* Received allo-hematopoietic stem cell transplantation therapy previously.
* Uncontrolled conditions or unwillingness or inability to follow the procedures required in the protocol;
* Received CAR T-cell or other genetically-modified T-cell therapy previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2028-08-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 months
  Objective response rate (ORR) in 3 month in relapsed and refractory (R/R) mantle cell lymphoma (MCL) subjects

SECONDARY OUTCOMES:
Complete response rate (CRR) | 3 months
  Complete response rate (CRR) in 3 month in relapsed and refractory (R/R) mantle cell lymphoma (MCL) subjects
The best objective response rate | 3 months
  The best objective response rate in 3 month in relapsed and refractory (R/R) mantle cell lymphoma (MCL) subjects
The best complete response rate | 3 months
  The best complete response rate in 3 month in relapsed and refractory (R/R) mantle cell lymphoma (MCL) subjects
Number of participants with adverse events (AEs) | Up to 24 months after JWCAR029 infusion
  Number of participants with adverse events
Type of adverse events (AEs) | Up to 24 months after JWCAR029 infusion
  Type of adverse events
Severity of adverse events(AEs) | Up to 24 months after JWCAR029 infusion
  Severity of adverse events
Number of participants with laboratory abnormalities | Up to 24 months after JWCAR029 infusion
  Number of participants with laboratory abnormalities
Type of laboratory abnormalities | Up to 24 months after JWCAR029 infusion
  Type of laboratory abnormalities
Severity of laboratory abnormalities | Up to 24 months after JWCAR029 infusion
  Severity of laboratory abnormalities
Duration of response (DOR) | Up to 24 months after JWCAR029 infusion
  Time from first response(PR or CR) to disease progression or death from any cause
Duration of complete remission (DoCR) | Up to 24 months after JWCAR029 infusion
  Time from complete response (CR) to disease progression or death from any cause
Duration of partial remission (DoPR) | Up to 24 months after JWCAR029 infusion
  Time from partial response (PR) to disease progression or death from any cause.
Time to response (TTR) | Up to 24 months after JWCAR029 infusion
  Time from JWCAR029 infusion to first documentation of complete response (CR) or partial response (PR)
Time to complete response (TTCR) | Up to 24 months after JWCAR029 infusion
  Time from JWCAR029 infusion to first documentation of complete response (CR)
Cmax of JWCAR029 | Up to 1 year after JWCAR029 infusion
  Maximum observed concentration of JWCAR029 in peripheral blood
Tmax of JWCAR029: | Up to 1 year after JWCAR029 infusion
  Time to maximum concentration of JWCAR029 in the peripheral blood
AUC of JWCAR029: | Up to 1 year after JWCAR029 infusion
  Area under the concentration vs time curve of JWCAR029 in the peripheral blood
Progression-free survival (PFS) | Up to 2 year after JWCAR029 infusion
  Progression-free survival
Overall survival (OS) | Up to 5 year after JWCAR029 infusion
  Overall survival
Anti-therapeutic JWCAR029 antibody | Up to 2 year after JWCAR029 infusion
  Anti-therapeutic JWCAR029 antibody
Changes of T cell counts | Up to 2 year after JWCAR029 infusion
  Changes of T cell counts
Changes of Subgroups of T cell | Up to 2 year after JWCAR029 infusion
  Changes of Subgroups of T cell
Changes of serum cytokines | Up to 2 year after JWCAR029 infusion
  Changes of serum cytokines
CD19 expression in tumor biopsy samples | Up to 2 year after JWCAR029 infusion
  CD19 expression in tumor biopsy samples
Changes in inflammatory biomarkers such as CRP | Up to 2 year after JWCAR029 infusion
  Changes in inflammatory biomarkers such as CRP
Changes in inflammatory biomarkers such as ferritin | Up to 2 year after JWCAR029 infusion
  Changes in inflammatory biomarkers such as CRP

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Consonancy Hospital, Fuzhou, Fujiang
  - Guangdong Province people hospital, Guanzhou, Guangdong
  - Henan Province Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province People Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Institute of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang province Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie Y, Zhou K, Li L, Liang A, Mei H, Zou D, Li W, Jin J, Jin Z, Jing HM, Yang H, Chen T, Huang H, He P, Cao J, Zhu J, Song Y, Xia Z, Gu YE, Zang Y, Zhou Z, Tian ZZ. Phase 2 Study of Relmacabtagene Autoleucel (CD19 CAR-T) for Relapsed/Refractory Mantle Cell Lymphoma in Chinese Adults. Blood Adv. 2025 Aug 14:bloodadvances.2024015763. doi: 10.1182/bloodadvances.2024015763. Online ahead of print. PMID 40811825